CLINICAL TRIAL: NCT03217630
Title: A Cohort Study of Ultrasound Evaluation of Gastric Emptying in Diabetic Patients: a Comparison With Non-diabetic Controls
Brief Title: Ultrasound Evaluation of Gastric Emptying in Diabetic Patients: a Comparison With Non-diabetic Controls
Status: Completed | Type: Observational
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Chunling Jiang, Professor, West China Hospital
Other Study IDs: 2017-141, 2018-56
Record Dates: First submitted 2017-07-09; First posted 2017-07-14 (Actual); Last update posted 2019-04-10 (Actual); Status verified 2019-04

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Diabetic patients
  Interventions: Other: Fasting 2 h after clear liquid or 6h after a light meal
- Non-diabetic patients
  Interventions: Other: Fasting 2 h after clear liquid or 6h after a light meal

INTERVENTIONS:
Other: Fasting 2 h after clear liquid or 6h after a light meal — The fasting time for all patients is 2 h after clear liquid or 6h after a light meal, then gastric ultrasound examination is performed.

SUMMARY:
This is a prospective cohort study. The main objective is to compare the prevalence of a "full stomach" using gastric ultrasound technique, in elective surgical patients with diabetes mellitus compared to non-diabetic controls following the present fasting guidelines (2 h after clear liquid and 6h after a light meal). For patients with a full stomach or intermediate stomach, an consecutive ultrasound scan is performed every 10 min,until empty stomachstomach contents are detected to determine the mean gastric emptying time for clear liquid and light meal, and to investigate the risk factors for delayed stomach emptying in diabetic patients by logistic regression analysis .

ELIGIBILITY:
Inclusion Criteria:

* diabetes (two fasting plasma glucose concentration≥7mmol/L or casual plasma glucose concentration≥11.1mmol/L);
* age≥18 yr; ASA physical status I-III;
* body mass index <35kg/m2;
* who are admitted to the surgical department;
* who are able to understand the rationale of the study and provide informed consent.

Exclusion Criteria:

* pregnancy;
* a history of upper gastrointestinal disease or previous surgery on the oesophagus, stomach or upper abdomen;
* documented abnormalities of the upper gastrointestinal tract such as gastric tumors;
* recent upper gastrointestinal bleeding (within the preceding 1 month);
* taking medicines that may delay gastric emptying(e.g., anticholinergic agents).
* hypothyroidism.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Study participants will be diabetic and non-diabetic patients who are admitted to the surgical department and scheduled to undergo elective surgical procedures. 100 participants will be recruited in total.
Sampling Method: Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Prevalence of full stomach | one day
  The frequency of a "full stomach" in the diabetic population compared to a non-diabetic control population at 2h after ingesting clear liquid or 6h after light meal.

SECONDARY OUTCOMES:
Mean gastric emptying time of clear liquid and light meal | one day
  The mean gastric emptying time of clear liquid and light meal in both diabetic and non-diabetic population.

OTHER OUTCOMES:
Risk factors of delayed stomach empty in diabetic patients | one day
  Correlation between the latest fast, postprandial plasma glucose concentration, hemoglobin A1c level and the diabetes complications ( peripheral neuropathy, cardiovascular autonomic neuropathy, diabetic nephropathy,and diabetes mellitus-related eye disease (including diabetic retinopathy, macular edema, rubeosis iridis, vitreous hemorrhage and diabetic related-visual injury)) with delayed stomach empty

CONTACTS AND LOCATIONS:
Overall Officials: Chunling Jiang, Principal Investigator — West China Hospital
Locations (1):
- West China Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zhou L, Yang Y, Yang L, Cao W, Jing H, Xu Y, Jiang X, Xu D, Xiao Q, Jiang C, Bo L. Point-of-care ultrasound defines gastric content in elective surgical patients with type 2 diabetes mellitus: a prospective cohort study. BMC Anesthesiol. 2019 Oct 10;19(1):179. doi: 10.1186/s12871-019-0848-x. PMID 31601180